CLINICAL TRIAL: NCT01640587
Title: Randomized Open-label Trial of Comparison Between DHA-Piperaquine and Mefloquine Artesunate Combinations 3 Day-regimens for the Treatment of Uncomplicated Plasmodium Falciparum Malaria on the Thai-Myanmar Border (RDM)
Brief Title: Compare the Effectiveness Between Existing Treatment and New Treatment
Acronym: RDM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No adequate malaria patient
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMRU1201
Record Dates: First submitted 2012-07-11; First posted 2012-07-13 (Estimated); Last update posted 2023-01-10 (Actual); Status verified 2017-06

CONDITIONS: P. Falciparum Malaria
Keywords: Uncomplicated falciparum infection; Mefloquine-artesunate; Dihydroartemisinin-piperaquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DP (Experimental): 2.4 mg/kg dihydroartemisinin AND 20 mg/kg piperaquine once daily on Days 0, 1 and 2
  Interventions: Drug: Dihydroartemisinin-Piperaquine
- MAS3 (Active Comparator): 4mg/kg artesunate AND 8 mg/kg mefloquine once daily on Days 0, 1 and 2
  Interventions: Drug: Mefloquine+Artesunate

INTERVENTIONS:
Drug: Mefloquine+Artesunate — One tablet of artesunate contains 40mg (Guilin Pharmaceutical Company, PRC). One tablet of mefloquine contains 250 mg mefloquine (Eloquine® (Medochemie Ltd., Cyprus) Standard three days regimen of artesunate-mefloquine given as 4mg/kg artesunate/day and 8 mg/kg of mefloquine/day on Days 0, 1 and 2
  Other Names: Eloquine®
  Arms: MAS3
Drug: Dihydroartemisinin-Piperaquine — DHA-Piperaquine (Duo-Cotecxin® Beijing Holley-Cotec Pharmaceuticals Co., Ltd, China) One tablet contains 40mg of dihydroartemisinin and 320 mg piperaquine. A weight-based regimen containing 2.4 mg/kg DHA and 20 mg/kg PPQ once daily for 3 days
  Other Names: Duo-Cotecxin®
  Arms: DP

SUMMARY:
In camps for displaced persons located along the Thai-Myanmar border, mefloquine and artesunate combination therapy has been used since 1992. In vivo efficacy of a 3 day regimen of mefloquine + artesunate (MAS3) has been monitored regularly since its introduction in 1992. In 2009 Carrara et al summarised the in vivo PCR-adjusted cure rates at Day 42 and Day 63 in patients treated with MAS3 between 1995 and 2005, as well as the in-vitro parasite susceptibility to MAS3 during that same period, and the changes in pfmdr1 copy numbers.The proportion of patients with parasitaemia persisting on day-2 increased significantly from 4.5% before 2001 to 21.9% after 2002 (p<0.001). Delayed parasite clearance was associated with increased risk of developing gametocytaemia (AOR = 2.29; 95% CI, 2.00-2.69, p = 0.002). MAS3 efficacy declined slightly but significantly (Hazards ratio 1.13; 95% CI, 1.07-1.19, p<0.001), although efficacy in 2007 remained well within acceptable limits: 96.5% (95% CI, 91.0-98.7). The proportion of infections caused by parasites with increased pfmdr1 copy number rose from 30% (12/40) in 1996 to 53% (24/45) in 2006 (p = 0.012, test for trend).

Evidence of reduced susceptibility to artemisinins in Western Cambodia was first reported in January 2007. Artemisinin resistance was manifest by a marked slowing of parasite clearance. A more recent analysis of parasite clearance data collected prospectively in patients with uncomplicated hyperparasitaemic malaria has shown a progressive decline in parasite clearance rates over the last decade suggesting a decline following the same trajectory as in Western Cambodia but with a time lag of a few years.

Surveillance data collected in 2011 have shown a dramatic and worrying decline in efficacy of MAS3, albeit in a small number of patients. This decline in efficacy of mefloquine + artesunate is likely to be attributable to reduced parasite susceptibility to mefloquine. The other fixed dose combinations available dihydroartemisinin-piperaquine (DP) is the best option to replace mefloquine-artesunate since it is thought that it remains effective in the presence of high pfmdr1 copy numbers. In addition DP is administered once daily and needs no special dietary modification to ensure adequate absorption.

In this study it is hypothesised that efficacy of DP (estimated to be 95%) will be significantly higher than that of MAS3 (estimated to be 65%), therefore the investigators propose to conduct a randomised controlled trial between DP and MAS3 for the treatment of P.falciparum.

DETAILED DESCRIPTION:
In camps for displaced persons located along the Thai-Myanmar border, mefloquine and artesunate combination therapy has been used since 1992. It was studied first in trials, but by 1994 it became the first line treatment for all uncomplicated P. falciparum malaria episodes in the non-pregnant population. In vivo efficacy of a 3 day regimen of mefloquine+ artesunate (MAS3) has been monitored regularly since its introduction in 1992. In 2009 Carrara et al summarised the in vivo PCR-adjusted cure rates at Day 42 and Day 63 in patients treated with MAS3 between 1995 and 2005, as well as the in-vitro parasite susceptibility to MAS3 during that same period, and the changes in pfmdr1 copy numbers.The proportion of patients with parasitaemia persisting on day-2 increased significantly from 4.5% before 2001 to 21.9% after 2002 (p<0.001). Delayed parasite clearance was associated with increased risk of developing gametocytaemia (AOR = 2.29; 95% CI, 2.00-2.69, p = 0.002). MAS3 efficacy declined slightly but significantly (Hazards ratio 1.13; 95% CI, 1.07-1.19, p<0.001), although efficacy in 2007 remained well within acceptable limits: 96.5% (95% CI, 91.0-98.7). The proportion of infections caused by parasites with increased pfmdr1 copy number rose from 30% (12/40) in 1996 to 53% (24/45) in 2006 (p = 0.012, test for trend).

Evidence of reduced susceptibility to artemisinins in Western Cambodia was first reported in January 2007. Artemisinin resistance was manifest by a marked slowing of parasite clearance. In Pailin, Cambodia, the median parasite clearance time was 84 hours compared to 48 hours on the Thai side of the international border with Myanmar following either 2 mg/kg of artesunate (AS) alone for 7 days or 4 mg/kg AS for 3 days plus 25 mg/kg of mefloquine at both locations. A more recent analysis of parasite clearance data collected prospectively in patients with uncomplicated hyperparasitaemic malaria has shown a progressive decline in parasite clearance rates over the last decade suggesting a decline following the same trajectory as in Western Cambodia but with a time lag of a few years.

Clinic experience data collected in 2011 have shown a steady decline in efficacy of MAS3, albeit in a small number of patients. We have observed this trend over the past 10 years. It appears to be related to the increased copies of the gene Pfmdr1 in adult males. The PCR corrected efficacy in 43 patients was 47.0% (95% CI 27.0-64.7), well below the 90% threshold at which WHO recommends changing to an alternative treatment. This decline in efficacy of mefloquine + artesunate is likely to be attributable to reduced parasite susceptibility to mefloquine. The other fixed dose combinations available dihydroartemisinin-piperaquine (DP) is the best option to replace mefloquine-artesunate since it is thought that it remains effective in the presence of high pfmdr1 copy numbers. In addition DP is administered once daily and needs no special dietary modification to ensure adequate absorption.

However other groups in the area have documented a good efficacy of MAS3. In other words we think there is a decline in efficacy but we do not feel confident to say what the magnitude of this drop is. Changing policy is a difficult task and we need more and stronger evidence of the current efficacy of MAS3. The best design to avoid selection bias is to do an adequately powered randomized control trial and we would like to compare MAS3 with the next generation ACT: DP. We have already conducted studies with DP and we know it is safe and effective. In laboratory studies we found that this treatment (DP) is more effective against P.falciparum when it exhibits resistance to mefloquine via increased expression of the Pfmdr1 gene. We think it is timely to compare MAS3 and DP again and carefully monitor for the treatment response in patients with signs of mefloquine resistant parasites. Therefore, we propose a study to evaluate in an adequately powered RCT MAS3 (the current national policy for Thailand and routinely use along the border) to a potential replacement, DP.

Due to a lack of malaria patients at clinics, the trial was terminated. There will be no further analysis and or publication of the results.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 5 years
* Symptomatic of malaria infection, i.e. history of fever or presence of fever >37.5°c.
* microscopically confirmed asexual stages of Plasmodium falciparum ≥ 5/500 wbc (may be mixed with non- P.falciparum species) .
* Written informed consent given to participate in the trial.
* Participant or parent/guardian is willing and able to give informed consent for participation in the study.
* Participant or guardian is able to understand and participant can complete the study requirements

Exclusion Criteria:

* Pregnancy or lactation (urine test for β HCG to be performed on any woman of child bearing age unless menstruating).
* P.falciparum asexual stage parasitaemia greater than or equal to 4% red blood cells (175 000/µL).
* Signs or symptoms indicative of severe malaria:

  * Impaired consciousness
  * Severe anaemia (Hct<15%)
  * Bleeding disorder -evidenced by epistaxis, bleeding gums, frank haematuria, bleeding from venepuncture sites.
  * Respiratory distress
  * Severe jaundice
* Patients who received any P. falciparum treatment within 2 months
* Known hypersensitivity to artemisinins - defined as history of erythroderma/ other severe cutaneous reaction, angioedema or anaphylaxis.
* History of epilepsy and other neurological disorders
* Splenectomy

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03-30 (Actual)

PRIMARY OUTCOMES:
PCR adjusted adequate clinical and parasitological response | Day 63
  Day 63 PCR adjusted adequate clinical and parasitological response (ACPR) in both DP3 arm and MAS3 arm

SECONDARY OUTCOMES:
PCR adjusted adequate clinical and parasitological response | Day 42
  Day 42 PCR adjusted adequate clinical and parasitological response (ACPR) in both DP3 arm and MAS3 arm
Proportion of aparasitaemic | Day 3
  Proportion of aparasitaemic patients on day 3 in both DP3 arm and MAS3 arm

CONTACTS AND LOCATIONS:
Overall Officials: Francois Nosten, MD, Principal Investigator — University of Oxford
Locations (1):
- Shoklo Malaria Research Unit, Mae Sot, Changwat Tak, Thailand